CLINICAL TRIAL: NCT07369167
Title: Neurophysiological, Kinematics and Functional Correlates of Goal-directed Action Observation and Execution in Children With Unilateral Cerebral Palsy
Brief Title: Neural Correlates of Goal-directed Action Observation and Execution in Children With Unilateral Cerebral Palsy
Acronym: EEG_AINCP
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Responsible Party: Principal Investigator, Giuseppina Sgandurra, Professor, IRCCS Fondazione Stella Maris
Other Study IDs: EEG_AINCP
Record Dates: First submitted 2026-01-16; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy (CP); Unilateral Cerebral Palsy; EEG; Action Observation
Keywords: Unilateral Cerebral Palsy; Mirror Neuron System; EEG; Mu rhythm; Sensorimotor; eye-tracker; wearable sensors; Action Observation; manual function; UCP
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: 40 children with Unilateral Cerebral Palsy (UCP), aged 5-15 years
- Control Group: 40 typically developing (TD) children, aged 5-15 years

SUMMARY:
Cerebral palsy (CP) is the most common childhood-onset motor disorder, with Unilateral Cerebral Palsy (UCP)- motor impairment predominantly impacting one side of the body-representing the most frequent form of CP. Among available rehabilitation programs, Action Observation Treatment (AOT) has gained increasing attention for its demonstrated effectiveness in improving manual motor function. AOT involves the systematic observation of goal-directed actions followed by their execution/imitation and is thought to leverage the mirror mechanism and its role in motor learning. Specifically, it relies on the neurophysiological principle that observing others' actions activates the same neural structures involved in executing those actions, reflecting the engagement of the mirror neuron system (MNS). In children with CP, the feasibility and effectiveness of AOT have been shown functionally (Sgandurra et al., 2013, Buchignani et al., 2019). However, despite its theoretical grounding in MNS functioning, the neurophysiological correlates of this system in children with CP remain less characterized, with only limited investigations using functional neuroimaging (e.g., Sgandurra et al., 2020) or neurophysiological methods such as electroencephalography (EEG; e.g., Demas et al., 2019).

This observational study aims to characterize the neurophysiological signatures of action execution and action observation in children aged 5-15 years with a diagnosis of UCP compared to a group of age-matched typically developing (TD) peers. To this end, non-invasive high-density EEG (hdEEG) will be used to quantify sensorimotor cortex modulation through mu-rhythm reactivity-specifically event-related desynchronization (ERD) and synchronization (ERS)-and its topographical distribution during an active visuo-motor task involving upper limbs. Mu-rhythm desynchronization (or suppression) over sensorimotor regions is a well-established marker of MNS engagement. A secondary objective is to examine the relationship between EEG measures and participants' attention, upper-limb kinematics, and manual motor function. To this purpose, participants will wear non-invasive wearable sensors to capture arm/hand kinematics, and attention will be monitored with a non-invasive eye-tracking system. Validated scales will be used to assess manual motor function.

Participants will take part in one single visit of about 1.5 hours. During the EEG acquisition session, children will wear a 128-channel EEG net and complete an active visuo-motor paradigm including the observation and execution of unimanual and bimanual goal-directed actions (e.g., reaching-grasping). In the observation condition, children will watch videos depicting these actions on a computer screen while refraining from movement. In the subsequent execution condition, they will interact themselves with the same objects as in the observation condition. Throughout the same session, children's attention/gaze will be tracked via eye-tracking, and upper-limb kinematics will be recorded using wearable inertial measurement unit (IMU) sensors. Before or after EEG acquisition, manual motor function will be assessed using two standardized scales: the Assisting Hand Assessment (AHA) and the Melbourne Assessment-2 (MA-2).

Data analysis will characterize the mu rhythm ERD topography and temporal dynamics during both action execution and action observation, within and between groups. Correlation analyses will explore associations between neurophysiological measures, gaze and attentional patterns, kinematic data, and motor assessments scores to elucidate how motor and attentional factors modulate sensorimotor cortical activation.

ELIGIBILITY:
Children with Unilateral Cerebral Palsy

Inclusion Criteria:

* Children with confirmed diagnosis of Unilateral Cerebral Palsy,
* Manual ability levels from I to III in the Manual Ability Classification System (MACS);
* Children's age from 5 to 15 years old.

Exclusion Criteria:

* Severe Upper Limb (UpL) impairment (MACS ≥ level IV: inability to grasp),
* UpL surgery within 12 months prior to study entry and botulinum toxin injection within 6 months prior to study entry,
* Severe comobordities,
* Severe cognitive disability, clinically assessed by the cognitive scales Wechsler, Preschool and Primary Scale of Intelligence (WPPSI-IV) or Wechsler Intelligence Scale for Children (WISC-IV or V).

Typically Developing children:

Inclusion Criteria

* 5 to 15 year-old children with typical development,
* No documented clinically relevant disorders

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with Unilateral CP (study group) - recruited at the IRCCS Fondazione Stella Maris Typically developing children (control group) - community sample
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Neurophysiological (EEG) data | 1 session - about 45 minutes
  - Mu-rhythm reactivity during the EEG action-observation task.
  Primary outcome measures will be the EEG mu rhythm modulation during the visuo-motor task performed by participants. The EEG mu rhythm suppression (or desynchronization) is an index of the human mirror neuron system activation over the sensorimotor cortex.
  Quantitative Spectral and time-frequency analyses will be performed to assess mu-rhythm suppression in response to executed and observed goal-directed actions.
  Mu rhythm event-related desynchronization/synchronization (ERD/ERS) patterns will be examined across scalp regions (primary region of interest: central and parietal sites) and conditions (observation, execution) and compared between groups (control group vs study group).

SECONDARY OUTCOMES:
Gaze behavior and Attentional engagement - during EEG session | 1 session: about 45 minutes (during EEG acquisition)
  Data on participants' gaze behavior and attentional engagement during EEG recording will be obtained from the eye tracking system. Analyses will focus on eye movements, stimulus fixation duration, and saccades during video observation. Eye-tracking measures will be correlated with EEG indices and compared between groups.
Kinematic data - during EEG session | 1 session: about 45 minutes (during EEG acquisition)
  Data from IMU wearable sensors will be acquired during EEG acquisition. Quantitative parameters for kinematics (i.e., position/trajectories, time, speed); dynamics (acceleration, forces); performance (jerk, accuracy, frequency and amplitude of movement) and symmetry and coordination indexes will be analyzed. These data will be correlated with EEG data and compared between groups.
Score of Assisting Hand Assessment (AHA) | 1 session: about 25-30 minutes (before or after EEG session)
  The AHA is a standardized assessment tool to measure the assisting hand performance in children with UCP. It can be used for children aged between 18 months and 18 years, with playful sessions made of semi-structured activities calibrated on different ages (different board games), and lasts approximately 25-30 minutes. The videotaped assessment is subsequently scored by a certified AHA examiner.
Score of the Melbourne Assessment 2 (MA-2) | 1 session: about 15 minutes (before or after EEG session)
  The MA-2 is a valid and reliable criterion-referenced test for evaluating upper limb movement quality in children with a neurological impairment aged 2.5 to 15 years. It consists of 14 unimanually tested items including reach, pointing, manipulation, grasp, release, and pro-/supination. Only the affected hand will be tested and it lasts approximately 15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppina Sgandurra, MD, PhD, Principal Investigator — IRCCS Fondazione Stella Maris
Locations (1):
- IRCCS Fondazione Stella Maris, Calambrone, Pisa, Italy

REFERENCES:
- [Background] Demas J, Bourguignon M, Perivier M, De Tiege X, Dinomais M, Van Bogaert P. Mu rhythm: State of the art with special focus on cerebral palsy. Ann Phys Rehabil Med. 2020 Oct;63(5):439-446. doi: 10.1016/j.rehab.2019.06.007. Epub 2019 Jul 9. PMID 31299375
- [Background] Buchignani B, Beani E, Pomeroy V, Iacono O, Sicola E, Perazza S, Bieber E, Feys H, Klingels K, Cioni G, Sgandurra G. Action observation training for rehabilitation in brain injuries: a systematic review and meta-analysis. BMC Neurol. 2019 Dec 27;19(1):344. doi: 10.1186/s12883-019-1533-x. PMID 31881854
- [Background] Sgandurra G, Ferrari A, Cossu G, Guzzetta A, Fogassi L, Cioni G. Randomized trial of observation and execution of upper extremity actions versus action alone in children with unilateral cerebral palsy. Neurorehabil Neural Repair. 2013 Nov-Dec;27(9):808-15. doi: 10.1177/1545968313497101. Epub 2013 Jul 25. PMID 23886886
- [Background] Sgandurra G, Biagi L, Fogassi L, Ferrari A, Sicola E, Guzzetta A, Tosetti M, Cioni G. Reorganization of action observation and sensory-motor networks after action observation therapy in children with congenital hemiplegia: A pilot study. Dev Neurobiol. 2020 Sep;80(9-10):351-360. doi: 10.1002/dneu.22783. Epub 2020 Oct 28. PMID 32986904